CLINICAL TRIAL: NCT05016050
Title: A Real-World Evidence, Single-Arm, Open-Label Study Evaluating the Safety and Efficacy of HPDT-DA-013 Digital Therapeutic in the Treatment of Major Depressive Disorder(MDD)and Generalized Anxiety Disorder(GAD)
Brief Title: Digital Therapeutic for Major Depressive Disorder (MDD) and Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happify Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HPY-HPDT-DA-013-RWE-01
Record Dates: First submitted 2021-08-16; First posted 2021-08-23 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: Major Depressive Disorder; Generalized Anxiety Disorder
Keywords: depression; anxiety
MeSH Terms: conditions — Depressive Disorder, Major; Generalized Anxiety Disorder; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Digital therapeutic (Experimental): Use HPDT-DA-013 digital therapeutic for a period of 8-10 weeks.
  Interventions: Device: HPDT-DA-013

INTERVENTIONS:
Device: HPDT-DA-013 — Digital program with therapeutic interventions based on Cognitive Behavioral Therapy (CBT).

SUMMARY:
Participants with Major Depressive Disorder (MDD) or Generalized Anxiety Disorder (GAD) will use a prescribed digital therapeutic for 8-10 weeks, and will complete depression and anxiety measures during this time. After the treatment period, participants will be followed monthly for 12 months.

DETAILED DESCRIPTION:
This study aims to assess the safety and efficacy of HPDT-DA-013 digital therapeutic in adults ages 22 years and older with MDD or GAD. Participants access HPDT-DA-013 on their smart device or computer and complete treatment over a period of 8-10 weeks. During the treatment period, participants complete PHQ-9 and GAD-7 assessments, as well as safety and medication use questionnaires. After 8-10 weeks, participants will complete end-of-treatment assessments, and access to HPDT-DA-013 will be removed. Participants are then followed for a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Adults 22 years or older at the time of screening
2. Meets DSM-5 diagnostic criteria for Major Depressive Disorder or Generalized Anxiety Disorder
3. Access to and willingness to use computer equipment/smartphone compatible with the product platform over a functional network for the study duration
4. Currently residing in the United States

Key Exclusion Criteria:

1. Risk of suicide or has attempted suicide within 24 months of the screening visit
2. Moderate to severe substance use disorder
3. Current co-morbid psychiatric diagnosis including PTSD, Schizophrenia, Bipolar Disorder I or II, or Borderline Personality Disorder
4. Currently pregnant or planning to become pregnant during the treatment period

Note: Other protocol-defined inclusion/exclusion criteria applied.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire-9 (PHQ-9) | baseline to end of treatment (8-10 weeks)
  A 9-item self-report measure to assess symptoms of depression
Generalized Anxiety Disorder-7 (GAD-7) | baseline to end of treatment (8-10 weeks)
  A 7-item self-report measure to assess symptoms of anxiety

SECONDARY OUTCOMES:
PHQ-9 | Through study completion, average of 14 months
  A 9-item self-report measure to assess symptoms of depression
GAD-7 | Through study completion, average of 14 months
  A 7-item self-report measure to assess symptoms of anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vilardaga, Ph.D., Principal Investigator — Duke University
Locations (1):
- Happify Health (Remote), New York, New York, United States

IPD SHARING:
Plan to Share IPD: No